CLINICAL TRIAL: NCT00311753
Title: An Open-label Comparison of the Efficacy and Safety of the Low-molecular-weight Heparin (3000 U Anti-Xa Once Daily) With Unfractionated Heparin for the Prevention of Thromboembolic Complications in Acutely Ill Non-surgical Patients
Brief Title: Efficacy and Safety of Low-molecular Weight Heparin for Thromboprophylaxis in Acutely Ill Medical Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMEX839BDE02
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Embolism
Keywords: heparin, thromboprophylaxis, medical patients, acutely ill; Acutely ill non surgical patients; Immobilization
MeSH Terms: conditions — Embolism | interventions — certoparin; Heparin

ARMS (2):
- 1 (Experimental): Certoparin
  Interventions: Drug: Certoparin
- 2 (Active Comparator): Heparin
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Certoparin — Low-molecular-weight heparin, Certoparin (3000 U anti-Xa once daily) treatment period of 10 ± 2 days
  Arms: 1
Drug: Heparin — 7500 IU of unfractionated heparin administered twice daily during the treatment period of 10 ± 2 days
  Arms: 2

SUMMARY:
Acutely ill immobilized patients are at a high risk for thromboembolic events including deep venous thrombosis or pulmonary embolism. Unfractionated heparin (UFH) and low molecular weight heparins (LMWH) are thought to be effective in preventing thromboembolic events. This study is designed to provide efficacy and safety data for thromboprophylaxis with the LMWH certoparin in comparison to thromboprophylaxis with UFH in acutely ill non-surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization due to an acute non-surgical disease
* Significant decrease in mobility

Exclusion Criteria:

* Indication for anticoagulant or thrombolytic therapy
* Major surgical or invasive procedure within the 4 weeks that precede randomization
* Expected major surgical or invasive procedure (including spinal/peridural/epidural anesthesia or lumbar puncture) within the 2 weeks that follow the randomization
* Immobilization due to cast or fracture of lower extremity
* Immobilization lasting longer than 3 days in the period prior to randomization
* Heparin administration longer than 36 hours in the period prior to randomization
* Acute ischemic stroke

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The occurrence of thromboembolic events (proximal or distal DVT, PE or VTE related death) during treatment | 10 ± 2 days

SECONDARY OUTCOMES:
Thromboembolic events during follow-up period of 3 months | 90 days (± 7 days) after the end of the treatment
Safety endpoints occurring during the treatment period: Hemorrhage (major or minor), Thrombocytopenia, Symptomatic HIT type II, Induction of HIT-II specific antibodies | 10 ± 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Schellong SM, Haas S, Greinacher A, Schwanebeck U, Sieder C, Abletshauser C, Bramlage P, Riess H. An open-label comparison of the efficacy and safety of certoparin versus unfractionated heparin for the prevention of thromboembolic complications in acutely ill medical patients: CERTAIN. Expert Opin Pharmacother. 2010 Dec;11(18):2953-61. doi: 10.1517/14656566.2010.521498. Epub 2010 Oct 18. PMID 20950224